CLINICAL TRIAL: NCT02299219
Title: Teens Taking Charge: A Pilot Randomized Controlled Trial of an Online Self-Management and Transitional Care Program for Youth With Cancer
Brief Title: Teens Taking Charge: Managing Cancer Online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Université de Montréal (Other); Children's Hospital of Eastern Ontario (Other); St. Justine's Hospital (Other); Hamilton Health Sciences Corporation (Other); Institute for Clinical Evaluative Sciences (Other); McGill University (Other); McMaster University (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Clinician Scientist, Clinical Nurse Specialist/NP, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000045896
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: Adolescent; Internet Self-Management; Managing Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taking Charge Experimental Group (Experimental)
  Interventions: Behavioral: Taking Charge: Managing Cancer Online
- Control Group (Active Comparator)
  Interventions: Behavioral: Standard Medical Care and Cancer Resource Center

INTERVENTIONS:
Behavioral: Taking Charge: Managing Cancer Online — n addition to standard medical care, adolescents in the experimental group will receive the "Taking Charge: Managing Cancer Online" Internet self-management program. The intervention is a 12-module interactive multi-component treatment protocol that consists of Cancer-specific education, self-management strategies, and social support that is available in English and French.
  Arms: Taking Charge Experimental Group
Behavioral: Standard Medical Care and Cancer Resource Center — The control group is designed to control for the potential effects on outcomes of time, attention and computer use during the intervention. In addition to standard medical care, adolescents in the attention control group will be provided with access to a self-guided patient education study website, which will have two components: basic patient educational materials about Cancer ("Cancer Resource Centre") and online assessments.
  Arms: Control Group

SUMMARY:
Cancer is the most common potentially fatal disease of adolescence and the Internet represents an ideal means to deliver education, self-monitoring capabilities, and social support to enhance disease self-management by adolescents with cancer. While two interactive coping websites exist for young people with cancer, they are: (1) not interactive, (2) do not focus on helping youth gain skills for transition and independence, and (3) do not provide opportunities for meaningful social support. In summary, there is a crucial need to develop a comprehensive interactive Internet-based self-management program targeting AWC that is comprised of cancer education, self-management skills, and opportunities for social support, and that is cost-effective.

DETAILED DESCRIPTION:
Overall aim of this program of research is to develop and evaluate the "Teens Taking Charge: Managing Cancer Online" Internet intervention that will help AWC to better cope with their disease, improve their HRQL, and enhance readiness to transition to adult health care using a sequential phased approach. The first phase of this project has determined the self-management and transitional care needs of adolescents with cancer. The second phase consisted of website development and usability testing to ensure the website is easy to use and understand, and is efficient and satisfying to complete. Subsequently, we will assess the feasibility of the program and the outcomes from the use of the site in a randomized controlled trial (RCT) pilot study (Phase 3). This will inform the design and methods of the main trial, and will permit us to obtain estimates of treatment effects on AWC health outcomes to inform the calculation of an appropriate sample size for the future definitive RCT (Phase 4). The focus of this study is Phase 3. Phase 4 will be a multicentre randomized controlled trial to assess outcomes for teens that complete the intervention as compared to those of an attention control group.

ELIGIBILITY:
Inclusion Criteria:

* Parents and adolescents will be eligible to participate if the adolescents are:

  1. between 12-18 years of age
  2. diagnosed with cancer (at least 3 months from diagnosis)
  3. on active treatment
  4. able to speak and read English and/or French at a Grade 6 level

Exclusion Criteria:

* Adolescents will be excluded if they:

  1. have major cognitive impairments
  2. have reduced executive function that may impact their ability to understand and use the online program
  3. are terminal/palliative as determined by their oncologist Parents/caregivers are not eligible to participate in the study alone (without an adolescent)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Participant Accrual and Dropout Rates | 12 weeks
  These rates will be centrally tracked by the Clinical Research Project Coordinator
Fidelity (Any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures) | 12 weeks
  Any issues or difficulties encountered during implementation of the intervention, control strategy, or outcome measures will be tracked throughout the study by the Clinical Research Project Coordinator
Acceptability and Satisfaction with Intervention (rate their acceptability of and satisfaction with the intervention) | 12 weeks
  Post-treatment, adolescents with cancer and their parents in the intervention group will rate their acceptability of and satisfaction with the intervention
Engagement with Intervention (Google Analytics will be used to track patterns of website program usage) | 12 weeks
  Google Analytics will be used to track patterns of website program usage by adolescents with cancer and their parents

SECONDARY OUTCOMES:
Knowledge (Adolescent Cancer Knowledge Questionnaire) | 12 weeks
  Measured using the Adolescent Cancer Knowledge Questionnaire, a 15-item tool that assesses cancer-specific knowledge.
Self-Efficacy (Generalized Self-Efficacy-Sherer Scale) | 12 weeks
  Measured by the Generalized Self-Efficacy-Sherer Scale, a 12-item scale that requires adolescents to indicate their level of agreement with a series of statements about self-efficacy.
Treatment adherence (Medication Adherence Scale) | 12 weeks
  Measured with the Medication Adherence Scale, a 4-item scale for assessing self-reported adherence.
Physical Symptoms - Pain (short form Brief Pain Inventory (BPI) | 12 weeks
  Measured using the short form Brief Pain Inventory (BPI), a 15-item measure that includes scales for measuring pain intensity, impact of pain on functioning and well being, and pain interference.
Physical Symptoms - Fatigue (PedsQL Multidimensional Fatigue Module) | 12 weeks
  Measured using the PedsQL Multidimensional Fatigue Module, an 18-item scale with validated versions for child report (ages 8-12 years), teen report (ages 13-18 years), and parental report for children and teens.
Emotional symptoms (Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Measured using the Hospital Anxiety and Depression Scale (HADS), a 14-item measure for individuals aged >12 years, which can be completed within 2-5 minutes.
Social functioning (Perceived Social Support from Friends (PSS-Fr) Scale) | 12 weeks
  Measured with the Perceived Social Support from Friends (PSS-Fr) Scale, a 20-item scale that assesses the extent to which an individual perceives that their friends fulfill their needs for support.
Transition readiness (Cancer Transition Scales) | 12 weeks
  Measured with the Cancer Transition Scales, which include sub-scales for 'cancer worry' (6 items), 'self-management skills' (15 items), and 'expectations' (12 items).
Health Related Quality of Life (PedsQL Cancer Module) | 12 weeks
  measured with the PedsQL Cancer Module, a 27-item scale, which has validated versions for child, teen, and parental report, and the Health Utility Index [HUI].
Cost effectiveness (ascertaining direct health care costs and family out of pocket costs) | 12 weeks
  Measured by ascertaining direct health care costs and family out of pocket costs related to cancer care incurred over the 12-week study period using the Health Care Utilization form modified from the Ambulatory and Home Care Record84-90 as well as direct costs related to the online intervention technology, intervention training and personnel. Quality adjusted life years will be calculated using the HUI to determine the incremental cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Stinson, PhD, CPNP, Principal Investigator — The Hospital for Sick Children
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec